CLINICAL TRIAL: NCT05960851
Title: A Phase I, Participant- and Investigator-Blind, Single-center Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Multiple Doses of LY3871801 in Healthy Asian and Non-Asian Participants
Brief Title: A Study of LY3871801 in Healthy Asian and Non-Asian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18334; J3P-MC-FTAC (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3871801 (Part A) (Experimental): LY3871801 administered orally in Japanese and Non-Asian Participants.
  Interventions: Drug: LY3871801
- Placebo (Part A) (Placebo Comparator): Placebo administered orally in Japanese and Non-Asian Participants.
  Interventions: Drug: Placebo
- LY3871801 (Part B) (Experimental): LY3871801 administered orally in Chinese Participants.
  Interventions: Drug: LY3871801
- Placebo (Part B) (Placebo Comparator): Placebo administered orally in Chinese Participants.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3871801 — Administered orally.
  Arms: LY3871801 (Part A); LY3871801 (Part B)
Drug: Placebo — Administered orally.
  Arms: Placebo (Part A); Placebo (Part B)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3871801 when administered as multiple doses in Healthy Asian and Non-Asian Participants. The study will also evaluate the amount of LY3871801 that gets into the blood stream and how long it takes the body to get rid of it in these participants. The study will be conducted in two parts (A & B). The study will last up to approximately 24 days excluding the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Are Japanese, Chinese, or Non-Asian participants who are overtly healthy as determined by medical evaluation
* Have body weight of >/= 45 kilograms (kg) & a body mass index (BMI) in the range of 18.5 to 29.5 kilogram per square meter (kg/m²). The Japanese participants must have a body weight of 45 to 85 kg and a BMI of 18.0 to 29.5 kg/m²

Exclusion Criteria:

* Have known allergies to LY3871801, related compounds, or any components of the formulation, or history of significant atopy
* Have a significant history of or current cardiovascular or heart failure (based on New York Heart Association Functional Classification), respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs
* Are females who are lactating or have a positive pregnancy test at screening or Day 1
* Positive for drug or alcohol screen at screening or Day -1
* Smoke more than 10 cigarettes per day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Predose up to 24 days post dose
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3871801 | Predose on Day 1 up to postdose on Day 17
  PK: Cmax of LY3871801
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3871801 | Predose on Day 1 up to postdose on Day 17
  PK: AUC of LY3871801

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Altasciences Clinical Los Angeles, Inc, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No